CLINICAL TRIAL: NCT05074966
Title: A Phase III, Multicenter, Open-label, Randomized Study to Assess the Efficacy and Safety of mXELOX Plus Cetuximab Versus FOLFOX Plus Cetuximab in Chinese Patients With RAS and BRAF Wild-type Metastatic Colorectal Cancer
Brief Title: The Efficacy and Safety of Modified XELOX(mXELOX) Plus Cetuximab vs FOLFOX Plus Cetuximab in RAS and BRAF WT mCRC Pts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Deputy director of Internal Medicine, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mCRC-CLARIFY-2021
Record Dates: First submitted 2021-09-07; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: patients with RAS/BRAF wild type left-sided mCRC will be randomized to two groups, which are mXELOX plus cetuximab and FOLFOX plus cetuximab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mXELOX plus cetuximab (Experimental): Patients will receive the study drug after randomization, and those with effective efficacy evaluation (CR, PR or SD) will receive intravenous chemotherapy for up to 9 cycles, and then enter the maintenance treatment stage until PD, death, intolerable toxicity or withdrawal of informed consent (whichever occurs first)
  Cetuximab: 500 mg/m2, IV, d1, q2w; Oxaliplatin: 85 mg/m2, IV, d1,q2w; Capecitabine: 850 mg/m2, po, bid, d1-10, q2w;
  maintenance stage: Cetuximab: 500 mg/m2, IV, d1, q2w; Capecitabine: 850 mg/m2, po, bid, d1-10, q2w;
  Interventions: Drug: Experimental: mXELOX plus cetuximab
- FOLFOX plus cetuximab (Active Comparator): Patients will receive the study drug after randomization, and those with effective efficacy evaluation (CR, PR or SD) will receive intravenous chemotherapy for up to 9 cycles, and then enter the maintenance treatment stage until PD, death, intolerable toxicity or withdrawal of informed consent (whichever occurs first)
  Cetuximab：500 mg/m2, IV, d1, q2w Oxaliplatin： 85 mg/m2, IV d1, q2w; Leucovorin： 400 mg/m2 IV d1, q2w; 5-FU： 400 mg/m2 IV bolus on d1, then 1200 mg/m2/d x 2d(total 2400 mg/m2 over 46-48 hours) IV continuous infusion, q2w;
  maintenance stage: Cetuximab: 500 mg/m2, IV, d1, q2w; Leucovorin： 400 mg/m2 IV d1, q2w; 5-FU： 400 mg/m2 IV bolus on d1, then 1200 mg/m2/d x 2d(total 2400 mg/m2 over 46-48 hours) IV continuous infusion, q2w （Cetuximab combined with capecitabine can be used according to the patient's wishes and the nursing situation of intravenous catheterization）
  Interventions: Drug: Active Comparator: FOLFOX plus cetuximab

INTERVENTIONS:
Drug: Experimental: mXELOX plus cetuximab — Patients will receive the study drug after randomization, and those with effective efficacy evaluation (CR, PR or SD) will receive intravenous chemotherapy for up to 9 cycles, and then enter the maintenance treatment stage until PD, death, intolerable toxicity or withdrawal of informed consent (whichever occurs first)
  Cetuximab: 500 mg/m2, IV, d1, q2w; Oxaliplatin: 85 mg/m2, IV, d1,q2w; Capecitabine: 850 mg/m2, po, bid, q2w maintenance stage: Cetuximab: 500 mg/m2, IV, d1, q2w; Capecitabine: 850 mg/m2, po, bid, d1-10, q2w;
  Arms: mXELOX plus cetuximab
Drug: Active Comparator: FOLFOX plus cetuximab — Patients will receive the study drug after randomization, and those with effective efficacy evaluation (CR, PR or SD) will receive intravenous chemotherapy for up to 9 cycles, and then enter the maintenance treatment stage until PD, death, intolerable toxicity or withdrawal of informed consent (whichever occurs first)
  Oxaliplatin 85 mg/m2, IV d1; Leucovorin 400 mg/m2 IV d1; 5-FU 400 mg/m2 IV bolus on d1, then 1200 mg/m2/d x 2d(total 2400 mg/m2 over 46-48 hours) IV continuous infusion; q2w maintenance stage: Cetuximab: 500 mg/m2, IV, d1, q2w; Leucovorin： 400 mg/m2 IV d1, q2w; 5-FU： 400 mg/m2 IV bolus on d1, then 1200 mg/m2/d x 2d(total 2400 mg/m2 over 46-48hours) IV continuous infusion, q2w （Cetuximab combined with capecitabine can be used according to the patient's wishes and the nursing situation of intravenous catheterization）
  Arms: FOLFOX plus cetuximab

SUMMARY:
This is an open label, multicenter, randomized study in Chinese patients with RAS and BRAF wild-type mCRC. Participants were randomly assigned to cetuximab + FOLFOX (group A) and cetuximab + modified XELOX[mXELOX] (group B). All patients in groups A and B will be treated until progression of disease(PD), death, intolerable toxicity or withdrawal of informed consent, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent (ICF) prior to any study procedure.
* Patient must be ≥18 years of age, at the time of signing the informed consent.
* Patients who had histologically or cytologically confirmed RAS and BRAF wild-type, initially unresectable metastatic adenocarcinoma of the left-sided colon or rectum, excluding appendiceal or anal cancer.
* The patients were willing to receive FOLFOX /mXELOX plus cetuximab as the first-line treatment choice after the diagnosis of mCRC;
* At least one measurable metastatic lesion(s) as defined by RECIST version 1.1. Eastern Cooperative Oncology Group (ECOG) performance score was 0-1 or KPS score ≥ 80.
* Life expectancy of at least 12 weeks in the opinion of the investigator.
* Neutrophils ≥ 1.5 × 109 / L, platelet ≥ 75 × 109 / L and hemoglobin ≥ 9 g / dl; Total bilirubin ≤ 1.5 × upper limit of normal value (ULN); ASAT (SGOT) and / or ALAT (SGPT) ≤ 2.5 × UNL (≤5×ULN in case of liver metastases）； Alkaline phosphatase ≤ 2.5 × UNL (≤ 5 × ULN in case of liver metastases; ≤ 10× ULN in case of bone metastasis ）； LDH <1500 U/L; Creatinine clearance (calculated according to Cockcroft and Gault) >60 mL/min or serum creatinine ≤1.5×ULN.

Exclusion Criteria:

* Previously received chemotherapy for CRC, except for adjuvant therapy>9 months (chemotherapy with oxaliplatin) or >6 months (chemotherapy without oxaliplatin) before the start of the study
* Patients that has been treated with monoclonal antibody, VEGF pathway targeted therapy, EGFR pathway targeted therapy, or other signal transduction pathway inhibitors
* Radiotherapy, RFA, interventional therapy or surgery were performed within 28 days before the first medication (except for previous diagnostic biopsy)
* Other active malignant tumors, excluding those who have been disease free for more than 5 years or in situ cancer considered to have been cured by adequate treatment
* Brain metastasis or meningeal metastasis has been confirmed. Patients with neurological symptoms should receive brain CT / MRI examination to exclude metastasis
* Peripheral nerve disorder is above grade 1(NCI CTCAE Version 5 )
* Existing toxicity or unrecovered toxicity caused by previous treatment whose grade is above 2 according to CTCAE criteria(excluding anemia, alopecia, skin pigmentation)
* Ascites, pleural effusion or pericardial fluid requiring drainage in the past 4 weeks
* Patients who is suffering from intestinal obstruction, gastrointestinal bleeding, pulmonary fibrosis or interstitial pneumonia, renal failure, liver failure or cerebrovascular disease
* Diabetes was not controlled, defined as HbA1c > 7.5% after anti-diabetic drugs or hypertension was not controlled, defined as systolic / diastolic blood pressure > 140 / 90 mmHg after antihypertensive drug
* Myocardial infarction, severe/unstable angina, New York Heart Association (NYHA) class III or IV congestive heart failure in the past 12 months
* Patients who was allergic to any of the research drugs (cetuximab, 5-FU, oxaliplatin, capecitabine) in the past
* Deficiency in dihydropyrimidine dehydrogenase (DPD) as manifested by medical history of fluorouracil adverse reactions
* Known to be infected with human immunodeficiency virus (HIV), have acquired immunodeficiency syndrome (AIDS) related diseases, have active hepatitis B or hepatitis C
* Suffering from autoimmune diseases or history of organ transplantation requiring immunosuppressive therapy
* May increase the risk associated with participation in the study or administration of the study drug or mental illness that may interfere with the interpretation of research results
* Pregnant women (determined by serum human chorionic gonadotropin [hCG]) or lactating women, or plan to conceive during the treatment period, 2 months after cetuximab treatment and 6 months after capecitabine treatment. Women of childbearing age with positive or no pregnancy test at baseline. Women of childbearing age or sexually active men were not willing to use contraception during the study period, at least 2 months after cetuximab treatment and 6 months after capecitabine treatment. Postmenopausal women must be amenorrhea for at least 12 months to be considered infertile
* There are other serious diseases that the researchers believe patients cannot be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-06-24 (Estimated); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
median PFS | From Baseline to primary completion date, about 48 months
  from randomization to PD or death from any cause

SECONDARY OUTCOMES:
Number of Participants With Adverse Events（AEs） During Treatment Period | From Baseline to primary completion date, about 48 months
  AEs included serious Adverse Events(SAEs) and non-serious AEs. Causality to study treatment was determined by the investigator. Severity was graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Number of Participants With Hematology Abnormalities During Treatment Period | From Baseline to primary completion date, about 48 months
  Hematology abnormalities include leukocyte count, hemoglobin, blood platelet count and neutrophil count
Number of Participants With Electrolyte Abnormalities During Treatment Period | From Baseline to primary completion date, about 48 months
  Electrolyte abnormalities include K, Na, Ca and Mg
Number of Participants With Clinical chemistry Abnormalities During Treatment Period | From Baseline to primary completion date, about 48 months
  Clinical chemistry abnormalities include blood urea nitrogen(BUN), serum creatinine, alkaline phosphatase(ALP), aspartate aminotransferase(AST), alanine aminotransferase(ALT), etc.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CR29 (EORTC QLQ-CR29) | From Baseline to primary completion date, about 48 months
  Quality of life in patients with colorectal cancer is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) CR29. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit. The maximum and minimum values are 104 and 25 respectively, and the smaller the value, the better the quality of life.
Change From Baseline in 5-level EuroQol-5 Dimensions(EQ-5D-5L) | From Baseline to primary completion date, about 48 months
  Quality of life in patients with colorectal cancer is assessed using 5-level EuroQol-5 Dimensions(EQ-5D-5L). EQ-5D-5L comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises five dimensions(MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY / DEPRESSION) , each dimension now has five response levels: no problems, slight problems, moderate problems, severe problems, unable to /extreme problems. The EQ VAS records the respondent's overall current health on a vertical visual analogue scale, where the endpoints are labelled "The best health you can imagine" and "The worst health you can imagine". The EQ VAS provides a quantitative measure of the patient's perception of their overall health. One hundred means the best health you can imagine and Zero means the worst health you can imagine. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit.
objective response rate | From Baseline to primary completion date, about 48 months.
  The proportion of patients who acquired complete response and partial response during treatment.
Overall Survival OS | From Baseline to primary completion date, about 48 months
  from randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, Doctor, Principal Investigator — Cancer Hospital & Institute, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital & Institute, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No